CLINICAL TRIAL: NCT05678517
Title: Seven-year Outcomes Following Intensive Anti-vascular Endothelial Growth Factor Therapy in Patients With Exudative Age-related Macular Degeneration
Brief Title: Seven-year Outcomes Following Intensive Anti-VEGF Therapy in Wet AMD
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Papp András, Associate Professor, Semmelweis University
Other Study IDs: SE RKB 168/2022
Record Dates: First submitted 2022-12-16; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients with AMD
  Interventions: Drug: Anti-VEGF

INTERVENTIONS:
Drug: Anti-VEGF — intravitreal ranibizumab or intravitreal aflibercept

SUMMARY:
The aim of this study was to assess long-term benefits of intensive aflibercept and ranibizumab anti-VEGF therapy in patients with exudative AMD.

DETAILED DESCRIPTION:
This study was conducted at two clinical sites in Budapest, Hungary after the "Vascular Endothelial Growth Factor (VEGF) Trap-Eye: Investigation of Efficacy and Safety in Wet Age-Related Macular Degeneration (VIEW 2)" phase-3 multicenter, prospective, randomized, double blind clinical trial (ClinicalTrials.gov ID: NCT00637377).

Patients were treated with intravitreal anti-VEGF injections between 2008 and 2017. During the first 2 years in the framework of the VIEW 2 study, participants were randomized per protocol to intravitreal aflibercept or ranibizumab treatment arms and received injections according to the VIEW 2 study protocol.

This study focused on long-term outcomes that happened after the VIEW 2 study. After finishing the VIEW 2 study, patients returned to daily routine medical care and were followed under regular clinical care in real-life conditions and were treated with predominantly ranibizumab anti-VEGF injections (participants received interventions as part of routine medical care). Treatment was administered as needed according to the judgement of the physician. Retreatment criteria were based on visual acuity, signs of activity on optical coherence tomography (OCT) or indirect slit lamp biomicroscopy. Results at the end of the follow-up (year 7) were retrospectively analyzed.

ELIGIBILITY:
* Same as the original VIEW2 study (NCT00637377)
* Finished VIEW 2 study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Same as the original VIEW2 study (NCT00637377)
  * Patients who finished the VIEW 2 study
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
BCVA | At the end of follow-up (year 7)
  Best-corrected visual acuity
Geographic atrophy | At the end of follow-up (year 7)
  Change in size of geographic atrophy on fundus autofluorescence (FAF)
Retinal fluid | At the end of follow-up (year 7)
  Presence or absence of intra- or subretinal fluid on spectral-domain optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Number of injections | Over the course of the follow-up (7 years)
  Number of intravitreal anti-VEGF injections given
Adverse events | Over the course of the follow-up (7 years)
  Potential adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Andras Papp, MD, PhD, Principal Investigator — Semmelweis University
Locations (2):
- Hungary (2):
  - Department of Ophthalmology, Semmelweis University, Budapest
  - Department of Ophthalmology, Bajcsy-Zsilinszky Hospital, Budapest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lukacs R, Schneider M, Nagy ZZ, Sandor GL, Kaan K, Asztalos A, Enyedi L, Pek G, Barcsay G, Szabo A, Borbandy A, Kovacs I, Resch MD, Papp A. Seven-year outcomes following intensive anti-vascular endothelial growth factor therapy in patients with exudative age-related macular degeneration. BMC Ophthalmol. 2023 Mar 17;23(1):110. doi: 10.1186/s12886-023-02843-2. PMID 36932356